CLINICAL TRIAL: NCT01010932
Title: Evaluation of Dotarem-enhanced MRA Compared to Time-Of-Flight (TOF) MRA in the Diagnosis of Carotid and Vertebral Basilar Arterial Disease
Brief Title: Carotid and Vertebral Magnetic Resonance Angiography (MRA) Study Comparing Dotarem and Time Of Flight (TOF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-048
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Arterial Diseases
Keywords: carotid or vertebral artery disease; Contrast agent; MRA
MeSH Terms: conditions — Cerebral Arterial Diseases | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dotarem and TOF MRA (Experimental): Each subject will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem enhanced MRA.
  Interventions: Drug: Dotarem; Other: TOF MRA

INTERVENTIONS:
Drug: Dotarem — Each subject will receive one injection of Dotarem 0.2ml/kg
  Other Names: Gadoterate meglumine
Other: TOF MRA — Each subject will undergo a Time of Flight Magnetic Resonance Angiography (TOF MRA)

SUMMARY:
The study will evaluate the efficacy and safety of Dotarem enhanced MRA in patients suffering from carotid or vertebral arterial disease.

DETAILED DESCRIPTION:
Each subject will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem enhanced MRA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 18 years
* Strongly suspected of having carotid or vertebral arterial disease
* Scheduled (or to be scheduled) to undergo computed tomography angiography (CTA) examination

Exclusion Criteria:

* Known grade IV or V chronic kidney disease (GFR<30 mL/min/1.73m²)
* Contraindication to MRI
* Acute renal dysfunction within the 6 months preceding Dotarem®-enhanced MRA examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DESCHE, MD, Study Director — Guerbet
Locations (1):
- Guerbet LLC, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit: 21 Sep 2009. Last patient last visit: 18 Nov 2010. Location: radiology departments
Pre-assignment Details: A total of 222 patients fulfilling the eligibility criteria were enrolled, of which 200 patients received Dotarem and completed the study. Twenty-two patients did not receive Dotarem and were discontinued prematurely.
Groups:
- TOF MRA Followed by Dotarem-enhanced MRA: Each patient will undergo a Time Of Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem-enhanced MRA.
  Each patient will be scheduled to undergo CTA either before TOF MRA or after Dotarem-enhanced MRA. CTA will be used as standard of truth.
Period: Overall Study
Arm/Group | TOF MRA Followed by Dotarem-enhanced MRA
Started | 222
Completed | 200
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | TOF MRA Followed by Dotarem-enhanced MRA
Number analyzed (Participants) | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 108
  >=65 years | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 117
Region of Enrollment [Number; unit: participants]
  United States | 81
  Colombia | 35
  Argentina | 48
  Mexico | 18
  Korea, Republic of | 39
  Chile | 1

OUTCOME MEASURES:

1. Primary Outcome: Technical Failure Rate
Description: Rate of non-assessable arterial segments as measured by 3 independent readers in off-site evaluation of TOF-MRA and Dotarem-enhanced MRA (re-read DGD-44-060).
Time Frame: 2 - 28 days
Population: For 2 patients, MRA images were not analyzed because images were incomplete.
Measure: Number (95% Confidence Interval); unit: percentage of arterial segments
Units Other Than Participants: arterial segments
Groups:
- Dotarem-enhanced MRA: Patients benefiting from an MRA after Dotarem IV administration
- TOF MRA: Patients benefiting from an MRA with no contrast medium administration
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 198 | 198
Number analyzed (arterial segments) | 2772 | 2772
percentage of arterial segments
  Reader 1 | 4.65 [3.87 to 5.44] | 29.44 [27.74 to 31.13]
  Reader 2 | 1.77 [1.28 to 2.26] | 16.70 [15.31 to 18.09]
  Reader 3 | 2.20 [1.65 to 2.75] | 18.54 [17.10 to 19.99]

2. Primary Outcome: Sensitivity
Description: Rate of true stenotic segments (i.e. with stenosis >= 70%) of TOF and Dotarem-enhanced MRA evaluated by 3 independent off-site readers at the segment level, with CTA as standard of truth (re-read DGD-44-060).
Time Frame: 2-42 days
Population: For 3 patients, MRA images were not analyzed: 2 patients with incomplete images and 1 patient who did not undergo CTA procedure.
Measure: Number (95% Confidence Interval); unit: percentage of stenotic segments
Units Other Than Participants: number of arterial segments
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 197 | 197
Number analyzed (number of arterial segments) | 2686 | 2686
percentage of stenotic segments
  Reader 1 | 58.46 [46.48 to 70.44] | 53.85 [41.73 to 65.97]
  Reader 2 | 63.08 [51.34 to 74.81] | 63.08 [51.34 to 74.81]
  Reader 3 | 53.85 [41.73 to 65.97] | 49.23 [37.08 to 61.38]

3. Primary Outcome: Specificity
Description: Rate of true non-stenotic segments (i.e. without stenosis >= 70%) of TOF and Dotarem-enhanced MRA evaluated by 3 independent off-site readers at the segment level, with CTA as standard of truth (re-read DGD-44-060).
Time Frame: 2 - 42 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of non-stenotic segments
Units Other Than Participants: Number of arterial segments
Arm/Group | Dotarem-enhanced MRA | TOF MRA
Number analyzed (Participants) | 197 | 197
Number analyzed (Number of arterial segments) | 2686 | 2686
percentage of non-stenotic segments
  Reader 1 | 98.13 [97.61 to 98.65] | 85.43 [84.07 to 86.78]
  Reader 2 | 98.51 [98.05 to 98.98] | 90.39 [89.26 to 91.51]
  Reader 3 | 98.63 [98.18 to 99.07] | 90.42 [89.30 to 91.55]

ADVERSE EVENTS:
Time Frame: Adverse events were collected since the patient signing the patient consent form till the end of the last visits, maximum duration is 42 days.
Description: Adverse Events reported during the 24 hours following TOF, 24 hours following Dotarem-enhanced MRA and 24 hours following CTA and Adverse Events in discontinued patients without Dotarem administration are described. Participants at risk were subjects exposed to Dotarem administration.
Groups:
- Dotarem MRA: Patients benefiting from a MR angiography after an IV administration of Dotarem
- TOF MRA: Patients benefiting from a MR angiography with no contrast medium administration
- Computerized Tomography Angiography (CTA): Patients benefiting from a CT angiography with an IV injection of iodinated contrast medium
- Patients Discontinued Without Dotarem Administration: Patients withdrawn before administration of Dotarem whatever the reason
Arm/Group | Dotarem MRA | TOF MRA | Computerized Tomography Angiography (CTA) | Patients Discontinued Without Dotarem Administration
Serious Adverse Events (participants affected / at risk) | 1/200 | 0/200 | 2/200 | 1/22
Other Adverse Events (participants affected / at risk) | 12/200 | 0/200 | 7/200 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem MRA (N=200) | TOF MRA (N=200) | Computerized Tomography Angiography (CTA) (N=200) | Patients Discontinued Without Dotarem Administration (N=22)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not related to Dotarem administration
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not related to Dotarem administration
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — not related to Dotarem administration
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not related to Dotarem administration
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem MRA (N=200) | TOF MRA (N=200) | Computerized Tomography Angiography (CTA) (N=200) | Patients Discontinued Without Dotarem Administration (N=22)
Injection site hematoma (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutrophil Count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less